CLINICAL TRIAL: NCT06342778
Title: An Open-label, Randomized, Crossover, Two-period Study of the Comparative Pharmacokinetics and Bioequivalence of Doxylamine+Pyridoxine, 10 mg + 10 mg Enteric-soluble Film-coated Tablets (Valenta Pharm JSC, Russia) and Diclectin, 10 mg + 10 mg Delayed-release Tablets (Duchesnay Inc, Canada) Under Fed Conditions in Healthy Volunteers
Brief Title: Pharmacokinetics and Bioequivalence of Doxylamine+Pyridoxine and Diclectin Under Fed Conditions in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DIP-05-02-2023
Record Dates: First submitted 2024-03-11; First posted 2024-04-02 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Nausea
MeSH Terms: conditions — Nausea | interventions — dicyclomine, doxylamine, pyridoxine drug combination; Doxylamine; Pyridoxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT-sequence (Experimental): Group 1 (14 volunteers, RT sequence) will take 2 tablets of Diclectin in Period 1 and 2 tablets of Doxylamine + Pyridoxine in Period 2
  Interventions: Drug: Doxylamine + Pyridoxine; Drug: Diclectin
- TR-sequence (Active Comparator): Group 2 (14 volunteers, TR sequence) will take 2 tablets of Doxylamine + Pyridoxine in Period 1 and 2 tablets of Diclectin in Period 2
  Interventions: Drug: Doxylamine + Pyridoxine; Drug: Diclectin

INTERVENTIONS:
Drug: Doxylamine + Pyridoxine — A single dose of R or T drug in each of 2 periods of the study under fed conditions
  Other Names: Doxylamine + Pyridoxine, enteric soluble film-coated tablets
Drug: Diclectin — A single dose of R or T drug in each of 2 periods of the study under fed conditions
  Other Names: Doxylamine + Pyridoxine, Delayed-release Tablets

SUMMARY:
This study aims to evaluate pharmacokinetic profile and establish bioequivalence of the investigational drug Doxylamine + Pyridoxine, enteric-soluble, film-coated tablets, 10 mg + 10 mg (Valenta Pharm JSC, Russia) compared to the reference drug Diclectin, delayed-release tablets, 10 mg + 10 mg (registration certificate holder - Tzamal Bio-Pharma, Israel, manufacturer - Duchesnay Inc, Canada) in healthy volunteers under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and personally signed informed consent form by the heathy subject prior to initiation of any study procedures.
2. Women of childbearing potential (18 to 49 years inclusive).
3. Verified "healthy" status with no abnormalities detected based on clinical, laboratory, and instrumental examinations specified in the study protocol.
4. Blood pressure (BP) level: systolic blood pressure (SBP) from 100 to 139 mmHg, diastolic blood pressure (DBP) from 60 to 89 mmHg (inclusive).
5. Heart rate (HR) from 60 to 90 beats per min (inclusive).
6. Respiratory rate (RR) 12 to 18 breaths per min (inclusive).
7. Body temperature from 36 to 36.9°C (inclusive).
8. Body mass index (BMI) of 18.5 ≤ BMI ≤ 30 kg/m², with body weight ≥ 45 kg.
9. Consent to use adequate contraceptive methods throughout the study and for 30 days after completion of the study, negative pregnancy test.
10. Volunteers must demonstrate appropriate behavior and coherent speech.

Non-inclusion Criteria:

1. Positive allergic history.
2. History of hypersensitivity to the active ingridient and/or excipients of the study drugs.
3. A history of drug intolerance to the active ingridient and/or excipients of the study medications.
4. Chronic diseases of cardiovascular, lymphatic, respiratory, nervous, endocrine, digestive, musculoskeletal, integumentary, immune systems, as well as genitourinary apparatus and hematopoietic organs.
5. Clinically significant deviations from normal reference values for laboratory and diadnostic parameters based on local laboratory standarts.
6. History of gastrointestinal tract surgery (excluding appendectomy performed at least 1 year prior to screening).
7. Diseases/conditions that, in the investigator's judgement, may affect the absorption, distribution, metabolism, or excretion of study drugs.
8. Acute infectious diseases within 4 weeks prior to screening.
9. Use of medications with significant effects on hemodynamics or those affecting liver fuction (barbiturates, benzodiazepines, omeprazole, cimetidine, etc.) within 1 month prior to screening.
10. Regular use of medicatins within 3 weeks prir to screening or single-dose medication intake within 7 days prior to screening.
11. Blood or plasma donation within 3 months prior to the Screening Visit.
12. Use of hormonal contraceptives within 2 months prior to the Screening Visit.
13. Use of depot injections of any medications within 3 months prior to the Screening Visit.
14. Pregnancy or lactation period, positive pregnancy test.
15. Participation in another clinical trial less than 3 months prior to screening or concurrently with the present study.
16. Consumption of more than 10 units of alcohol (1 unit of alcohol is equivalent to 500 mL of beer, 200 mL of wine, or 50 mL of spirits) per week in the last month prior to inclusion in the study or history of alcoholism, drug abuse, or medicines abuse.
17. Smoking.
18. Positive blood test for antibodies to human immunodeficiency virus (HIV) types 1 and 2, antibodies to Treponema pallidum antigens, hepatitis B surface antigen (HBsAg), antibodies to hepatitis C virus antigens, rapid test (nasopharyngeal and/or oropharyngeal swab) for SARS-Cov-2 (COVID-19).
19. Clinically significant abnormalities on electrocardiogram (ECG).
20. Positive urinalysis for narcotics and potent drugs.
21. Positive breath alcohol vapor test.
22. Scheduling a hospital stay during the study period, for any reason other than hospitalization required by this protocol.
23. Inability or inability to comply with the requirements of the protocol, to follow the procedures prescribed by the protocol, to follow the diet, activity regime.
24. Observance of religious fasting or special diet (e.g., vegetarian, vegan).
25. Other conditions that, in the Investigator's judgement, may interfere with the volunteer's participation in the study or lead to early withdrawal, including lifestyle factors such as night shift work or extreme physical exertion.

Exclusion criteria

1. Refusal by the volunteer to continue participation in the study.
2. Failure of the volunteer to comply with study protocol requirements, including missed visits, unauthorized use of prohibited medications, or non-adherence to dietary and lifestyle restrictions.
3. Occurrence of safety-related issues during the study that endanger the subject (e.g. hypersensitivity reactions, etc.).
4. Volunteers included in the study in violation of the inclusion/non-inclusion criteria.
5. Volunteer developing a severe and/or serious adverse event during the study.
6. Missing collection of 2 or more consecutive blood samples, or 3 or more blood samples within a single period of pharmacokinetic part of the study.
7. Occurrence of vomiting/diarrhea within 24 h after administration of the study drug (the choice of time interval is based on the value of tmax parameter for doxylamine and pyridoxal-5-phosphate, not exceeding 7.2 ± 1.9 and 11.7 ± 5.3 h, respectively, according to the manufacturer of the reference drug).
8. Positive urine test for narcotics and potent drugs.
9. Positive breath alcohol vapor test.
10. A positive pregnancy test.
11. A positive test for SARS-Cov-2 (COVID-19);
12. Development of any new condition or situation that hinders protocol-defined procedures.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | From 0 to 72 hours (Day 1-4 and Day 15-18)
  Maximum plasma concentration (Cmax) of doxylamine and pyridoxal-5-phosphate
Pharmacokinetics - tmax | From 0 to 72 hours (Day 1-4 and Day 15-18)
  Time to reach Cmax (tmax) of doxylamine and pyridoxal-5-phosphate
Pharmacokinetics - AUC0-t | From 0 to 72 hours (Day 1-4 and Day 15-18)
  Area under the plasma concentration-time curve from time 0 to t (AUC0-t) of doxylamine and pyridoxal-5-phosphate
Pharmacokinetics - AUC0-inf | From 0 to 72 hours (Day 1-4 and Day 15-18)
  Area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf) of doxylamine and pyridoxal-5-phosphate
Pharmacokinetics - AUCextr | From 0 to 72 hours (Day 1-4 and Day 15-18)
  Extrapolated AUC of doxylamine and pyridoxal-5-phosphate, defined as (AUC0-inf - AUC0-t)/AUC0-inf
Pharmacokinetics - t1/2 | From 0 to 72 hours (Day 1-4 and Day 15-18)
  Elimination half-life (t1/2) of doxylamine and pyridoxal-5-phosphate
Pharmacokinetics - kel | From 0 to 72 hours (Day 1-4 and Day 15-18)
  Elimination constant (kel) of doxylamine and pyridoxal-5-phosphate
Pharmacokinetics - MRT | From 0 to 72 hours (Day 1-4 and Day 15-18)
  Mean residence time (MRT) of doxylamine and pyridoxal-5-phosphate
Bioequivalence - ratio of Cmax | From 0 to 72 hours (Day 1-4 and Day 15-18)
  Ratio of geometric mean Cmax for doxylamine and pyridoxal-5-phosphate after intake of R or T (with 90% confidence intervals)
Bioequivalence - ratio of AUC0-t | From 0 to 72 hours (Day 1-4 and Day 15-18)
  Ratio of geometric mean AUC0-t for doxylamine and pyridoxal-5-phosphate after intake of R or T (with 90% confidence intervals)
Bioequivalence - ratio of AUC0-inf | From 0 to 72 hours (Day 1-4 and Day 15-18)
  Ratio of geometric mean AUC0-inf for doxylamine and pyridoxal-5-phosphate after intake of R or T (with 90% confidence intervals)

SECONDARY OUTCOMES:
Adverse event type | From Day - 14 to Day 0 (screening) to Day 22 ± 1 (end of the study)
  Adverse events will be assessed by complaints, results of physical examination, results of heart rate and blood pressure assessment, results of respiratory rate assessment, body temperature, laboratory monitoring (clinical blood count, biochemical blood count, urinalysis), electrocardiography; adverse events will be classified in accordance to MedDRA.
Adverse event frequency | From Day - 14 to Day 0 (screening) to Day 22 ± 1 (end of the study)
  Number and frequency of adverse events registered during the study
Adverse event severety | From Day - 14 to Day 0 (screening) to Day 22 ± 1 (end of the study)
  Severity of adverse events registered during the study

CONTACTS AND LOCATIONS:
Locations (1):
- State budgetary health care institution Yaroslavl region "Clinical Hospital № 3", Yaroslavl, Russia

IPD SHARING:
Plan to Share IPD: No